CLINICAL TRIAL: NCT01814462
Title: Impact of CPAP Therapy in Obstructive Sleep Apnea on Parameters of Nocturnal Pulse Wave Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WI_ASIC+CPAP_121/2012
Record Dates: First submitted 2013-03-11; First posted 2013-03-20 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Pulse wave analysis
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6 months CPAP (Experimental): Application of continuous positive airway pressure (CPAP) therapy as established per routine clinical treatment. Home use of therapy for a period of 6 months.
  Interventions: Device: 6 months CPAP

INTERVENTIONS:
Device: 6 months CPAP

SUMMARY:
The present study aims to document and assess changes in single parameters of pulse wave analysis (ASI single parameters) as well as to evaluate ASI cardiovascular risk assessment before initiation of CPAP therapy and after 6 months of CPAP therapy in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repeated occurrence of apneas or reduced inspiratory air flow due to obstructions of the upper airways (hypopneas). These recurring events are accompanied by intermittent hypoxemia and sympathetic activation, leading to hemodynamic oscillations including relevant variations of pulse wave and blood pressure. Thus, OSA is associated with cardiovascular diseases and was identified as an independent risk factor for hypertension.

Direct effects of obstructive respiratory events (obstructive apneas and hypopneas) include changes of the peripheral pulse wave. The latter can easily be measured by finger plethysmography, e.g. by using established pulse oximeters. Certain pulse wave characteristics and their reaction towards obstructive respiratory events may provide information on cardiovascular function and thereby help in individual cardiovascular risk assessment.

Recently, Grote et al. published a concept for cardiovascular risk assessment based on pulse oximetry and pulse wave analysis ("ASI" - Grote et al. 2011, CHEST). The algorithm described herein is able to differentiate between high and low risk patients according to ESH/ESC risk classification (high risk = 4 and 5, low risk 1-3). To that end, oxygen saturation as measured by pulse oximetry, reductions in pulse wave amplitude, pulse rate accelerations, pulse propagation time and cardiorespiratory coupling are taken into account to calculate a quantitative total risk.

A successful OSA therapy applying positive airway pressure (e.g. CPAP) normalizes sleep-related breathing disturbances and thus counterbalances hemodynamic oscillations. This presumably results in reduced cardiovascular risk and should be detectable by measurable changes in pulse wave. This study aims to evaluate these effects by analyzing the single pulse wave parameters, which are part of the ASI algorithm. At the same time, established risk factors as well as the objective therapy outcome will be documented from the established sleep medicine viewpoint.

ELIGIBILITY:
Inclusion Criteria:

* Sleep-related breathing disorders with an apnea-hypopnea index ≥15/h and <30% central respiratory events (OSA patients)
* Stable optimal medication according to European Society of Cardiology guidelines (if applicable)

Exclusion Criteria:

* Prior exposure to positive airway pressure treatment
* Atrial fibrillation
* Facial anomalies or injuries inhibiting proper mask fit
* Pregnancy and/or lactation
* Acute life-threatening illness (e.g. instable angina pectoris, acute bronchial asthma, heart failure New York Heart Association stage IV, myocardial infarction, exacerbated Chronic obstructive pulmonary disease, malignant tumor requiring treatment)
* Drug or alcohol abuse
* Intake of hypnotics/sedatives
* Any medical, psychological or other condition impairing the patient's ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Change in pulse wave attenuation index | 6 months
  The pulse wave attenuation index represents the number of decreases of the pulse wave amplitude >10% and <30% compared with baseline (a moving median value of 20 samples surrounding the observed sample). This number is given as attenuations per hour. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.

SECONDARY OUTCOMES:
Change in mean pulse propagation time | 6 months
  The pulse propagation time represents the time interval between the systolic and dicrotic notch of the pulse wave form. The mean pulse propagation time of a complete recording is documented. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.
Change in mean respiration-related pulse oscillation | 6 months
  The respiration-related pulse oscillation is calculated by measuring the breathing-associated oscillation (respiratory sinus arrhythmia in the frequency band between 0.15 and 0.4 Hz) from the pulse rate signal in the time domain. The mean respiration-related pulse oscillation value of a complete recording is documented. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.
Change in pulse rate acceleration index | 6 months
  The pulse rate acceleration index represents the number of pulse rate increases ≥10% from baseline (a moving median value of 20 samples surrounding the observed sample). This number is given as increases per hour. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.
Change in hypoxia index | 6 months
  The hypoxia index represents the number of oxygen desaturation events per hour. A desaturation event is defined as a ≥2% drop of saturation of each sample compared with a 90 seconds time window of the upcoming SpO2 signal. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.
Change in ASI cardiovascular risk score | 6 months
  The ASI algorithm described by Grote et al. (2011) combines several single parameters from pulse wave analysis to calculate an overall cardiovascular risk score. The difference from baseline (without therapy) to 6 months (on CPAP therapy) is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Hospital, Solingen, Germany

REFERENCES:
- [Background] Grote L, Sommermeyer D, Zou D, Eder DN, Hedner J. Oximeter-based autonomic state indicator algorithm for cardiovascular risk assessment. Chest. 2011 Feb;139(2):253-259. doi: 10.1378/chest.09-3029. Epub 2010 Jul 29. PMID 20671056
- [Background] Lavie P, Herer P, Hoffstein V. Obstructive sleep apnoea syndrome as a risk factor for hypertension: population study. BMJ. 2000 Feb 19;320(7233):479-82. doi: 10.1136/bmj.320.7233.479. PMID 10678860
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Young T, Peppard P, Palta M, Hla KM, Finn L, Morgan B, Skatrud J. Population-based study of sleep-disordered breathing as a risk factor for hypertension. Arch Intern Med. 1997 Aug 11-25;157(15):1746-52. PMID 9250236
- [Background] Grote L, Ploch T, Heitmann J, Knaack L, Penzel T, Peter JH. Sleep-related breathing disorder is an independent risk factor for systemic hypertension. Am J Respir Crit Care Med. 1999 Dec;160(6):1875-82. doi: 10.1164/ajrccm.160.6.9811054. PMID 10588600
- [Background] Bixler EO, Vgontzas AN, Lin HM, Ten Have T, Leiby BE, Vela-Bueno A, Kales A. Association of hypertension and sleep-disordered breathing. Arch Intern Med. 2000 Aug 14-28;160(15):2289-95. doi: 10.1001/archinte.160.15.2289. PMID 10927725
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004 Aug;79(8):1036-46. doi: 10.4065/79.8.1036. PMID 15301332
- [Background] Peker Y, Hedner J, Norum J, Kraiczi H, Carlson J. Increased incidence of cardiovascular disease in middle-aged men with obstructive sleep apnea: a 7-year follow-up. Am J Respir Crit Care Med. 2002 Jul 15;166(2):159-65. doi: 10.1164/rccm.2105124. PMID 12119227
- [Background] O'Donnell CP, Ayuse T, King ED, Schwartz AR, Smith PL, Robotham JL. Airway obstruction during sleep increases blood pressure without arousal. J Appl Physiol (1985). 1996 Mar;80(3):773-81. doi: 10.1152/jappl.1996.80.3.773. PMID 8964736
- [Background] Davies RJ, Belt PJ, Roberts SJ, Ali NJ, Stradling JR. Arterial blood pressure responses to graded transient arousal from sleep in normal humans. J Appl Physiol (1985). 1993 Mar;74(3):1123-30. doi: 10.1152/jappl.1993.74.3.1123. PMID 8482650
- [Background] Buchner NJ, Sanner BM, Borgel J, Rump LC. Continuous positive airway pressure treatment of mild to moderate obstructive sleep apnea reduces cardiovascular risk. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1274-80. doi: 10.1164/rccm.200611-1588OC. Epub 2007 Aug 2. PMID 17673692
- [Background] Hui DS, Shang Q, Ko FW, Ng SS, Szeto CC, Ngai J, Tung AH, To KW, Chan TO, Yu CM. A prospective cohort study of the long-term effects of CPAP on carotid artery intima-media thickness in obstructive sleep apnea syndrome. Respir Res. 2012 Mar 16;13(1):22. doi: 10.1186/1465-9921-13-22. PMID 22424053